CLINICAL TRIAL: NCT00496093
Title: Safety, Tolerability and Immunogenicity of Pneumovax 23 (V110) in Healthy Adults in India
Brief Title: Safety, Tolerability and Immunogenicity of Pneumovax 23 in Healthy Adults in India (V110-011)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: V110-011; 2007_018
Record Dates: First submitted 2007-07-03; First posted 2007-07-04 (Estimated); Last update posted 2017-03-14 (Actual); Status verified 2017-03

CONDITIONS: Pneumococcal Infection
MeSH Terms: conditions — Pneumococcal Infections | interventions — Pneumococcal Vaccines; 2,4,5,4'-tetrachlorodiphenylsulfoxide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Pneumococcal Vaccine, Polyvalent (23-valent) (Experimental): Participants received one 0.5 mL dose of Pneumococcal Vaccine, Polyvalent (23-valent) by intramuscular (deltoid) injection on Day 1.
  Interventions: Biological: Pneumococcal Vaccine, Polyvalent (23-valent)

INTERVENTIONS:
Biological: Pneumococcal Vaccine, Polyvalent (23-valent)
  Other Names: V110; PNEUMOVAX™ 23

SUMMARY:
To describe the safety, tolerability and immunogenicity of pneumovax 23 (V110) in healthy adults in India.

DETAILED DESCRIPTION:
This was an open-label non-randomized study to assess the safety and immunogenicity of PNEUMOVAXTM 23 in healthy adults in India. The participants enrolled in this study were healthy Indian adults, 50 years of age or older, with no prior history of having received a pneumococcal vaccination (14-valent or 23-valent) and no prior history of Pneumococcal disease. All participants enrolled in the study received one 0.5 mL dose of PNEUMOVAXTM 23 by intramuscular (deltoid) injection on Day 1. Serum samples were obtained prior to vaccination on Day 1 and on Day 28 (+/-7 days) postvaccination. The duration of participation for each participant was approximately one month, with the study completion at the Day 28 postvaccination bleed and return of the Vaccination Report Card (VRC). Enrollment was completed within approximately 2 months. The last postvaccination blood sample was collected within 3 months of study initiation.

ELIGIBILITY:
Inclusion Criteria:

* Healthy indian adults of 50 years of age
* In good health; any underlying chronic illness must be documented to be in stable condition
* Signed and dated informed consent prior to receipt of the study vaccine

Exclusion Criteria:

* Functional or anatomic asplenia
* History of auto immune disease
* Hypersensitivity to any of the components of the study vaccine,including phenol
* Known or suspected immune dysfunction, including persons with congenital immunodeficiency
* Prior vaccination with any pneumococcal vaccine

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 133 (Actual)
Dates: Start 2005-10; Primary Completion 2006-01 (Actual); Study Completion 2006-01 (Actual)

PRIMARY OUTCOMES:
Percentage of subjects exhibiting a >= 2 fold increase in IGG antibody level from pre-vaccination to post-vaccination for both serotypes 1 and 6b | post-vaccination

SECONDARY OUTCOMES:
Any AE within 15 days after vaccination, with particular attention to injection site AE and fever | 15 days after vaccination

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

REFERENCES:
- Available data/document: CSR Synopsis — http://www.merck.com/clinical-trials/policies-perspectives.html